CLINICAL TRIAL: NCT05496920
Title: Assessing the Clinical Acceptability of Ultra-low Dose PET/CT and CT-less PET Using a Long Axial Field-of-view PET/CT System: a Single-centre, Single-blinded Method Agreement Study
Brief Title: Assessing Ultra-low Dose PET/CT and CT-less PET Using a Long Axial Field-of-view PET/CT System
Acronym: ULD-PET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-D0038
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: PET/CT
Keywords: PET/CT, low dose, long-axial field-of-view, extended field-of-view, total-body PET

STUDY DESIGN:
Intervention Model Description: Patients will receive first a standard of care PET/CT and then an additional low dose PET/CT. The low dose PET/CT will be reconstructed using a standard CT for attenuation correction (LD-PET/CT) and with a novel CT-less method using transmission data (ultra low dose ULD-PET/CT).
Masking Description: Scan reviewers will be masked to dose and scan reconstruction method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Patients will receive both a standard of care PET/CT and a low dose PET/CT
  Interventions: Diagnostic Test: FD-PET/CT; Diagnostic Test: LD-PET/CT

INTERVENTIONS:
Diagnostic Test: FD-PET/CT — Standard of care PET/CT with full dose (FD) of the radiopharmaceutical
Diagnostic Test: LD-PET/CT — Additional low dose PET/CT performed within protocol defined time frame LD-PET/CT with additional ultra-low dose CT-less reconstruction

SUMMARY:
Latest generation extended axial field-of-view (FOV) PET/CT systems offer the potential for substantial reductions in applied radiopharmaceutical necessary for a clinical scan. However, such low-dose examination protocols have yet to be robustly tested or demonstrated to be non-inferior. Furthermore, extended FOV scanners offer the potential for CT-less attenuation correction of the PET emission data, making clinically acceptable ultra-low dose examination protocols with radiation exposures of < 1 millisievert possible for the first time. The aim of this study is to demonstrate the clinical acceptability of such low and ultra-low dose scanning protocols in a head-to-head prospective study against a full-dose scan using a regular FOV system

DETAILED DESCRIPTION:
The first installation of a long-axial field-of-view (LAFOV) PET/CT system occurred in October 2020 at the department for nuclear medicine in Bern. This scanner along with recently introduced total-body scanners (TB-PET/CT) represent a substantial step forward in terms of nuclear medicine imaging technology. In conjunction with recent improvements in time-of-flight resolution and fully-digital detection technology, such systems offer surpassed sensitivity with improvements in image quality, lesion detection and diagnostic certainty. In contrast to LAFOV systems, standard axial field of view (SAFOV) scanners suffer from limited detection efficiency, where 90% of emitted photons go undetected owing to the ability to capture signal from only a small portion of the body (termed "bed position" or "bp").

However, while a number of studies are able to simulate lower applied radiopharmaceutical activities through the re-sampling of PET-sinogrammes or the rebinning of list-mode data, few studies adequately test the application of lower radiopharmaceutical activities, where limited data are available to justify the deviation from clinical routine. The clinical acceptability of such low-dose scans, in terms of lesion detection, image quality and lesion quantification is yet to be determined, which this study aims to address.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years) able to provide informed consent for inclusion, willing and able to undergo a PET/CT for the detection or staging of cancer.
* Individuals undergoing a PET/CT with 18F-FDG for the investigation of known or suspected NSCLC.
* Upper fasting plasma glucose levels of <8.3 mmol/L (<150 mg/dL) (as measured >30 mins prior to the administration of the radiopharmaceutical).

Exclusion Criteria:

* Patients who are unable to consent to a second study-specific examination
* Patients with claustrophobia requiring medication.
* Patients who commence active treatment of a cancer or other pathology between scans.
* Patients who have not fasted for > 4 hours prior to the study.
* Insulin dependent diabetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Intra-rater correlation coefficient | 2-6 weeks following scan
  ICC for Cancer Stage using the union for international cancer control (UICC) TNM (T= tumor, N= nodal stage, M = metastasis) System (8th Edition) for low dose positron emission and computed tomography (LD-PET/CT) exams compared to the standard of care (SOC) full-dose (FD)-PET/CT as assessed by a panel of physicians

SECONDARY OUTCOMES:
Intra-rater correlation coefficient | 2-6 weeks following scan
  ICC for ultra-low dose (ULD)-PET/CT compared to FD- and LD-PET/CT
Lesion uptake | 2-6 weeks following scan
  Composite outcome assessing lesion quantification in terms of peak standardised uptake value (SUVpeak), tumour to background (TBR), metabolic tumour volume (MTV) and tumour glycolytic activity (TLG) for ULD- and LD-PET/CT compared to the standard of care FD-PET/CT
Image quality | 2-6 weeks following scan
  Composite outcome assessing image quality in terms of tumour to background ratio (TBR) and signal to noise (SNR), defined as the reciprocal coefficient of variation (COV) for ULD- and LD-PET/CT compared to the standard of care FD-PET/CT
Subjective quality | 2-6 weeks following scan
  Image quality (subjective) as rated by five independent nuclear medicine physicians on a five-point Likert scale (1= unacceptable, 2=poor, 3=moderate, 4=good, 5=high) for ULD- and LD-PET/CT compared to the standard of care FD-PET/CT
Agreement | 2-6 weeks following scan
  Inter-reader agreement for the primary outcome (UICC cancer stage) shall be compared between LD and FD-PET/CT
Diagnostic accuracy | 2-6 weeks following scan
  Assessment of the positive predictive value (PPV) for LD- and FD-PET/CT for patients who undergo surgery or bronchoscopy and where histopathological confirmation of true positive (TP) and false positive (FP) findings are available

OTHER OUTCOMES:
Acceptability | 2-6 weeks following scan
  Additional outcome of interest: Patient and referrer acceptability of low-dose PET/CT examinations examined by means of a structured questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Axel O Rominger, MD, Study Chair — Inselspital
Locations (1):
- Inselspital, Universitätsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No